CLINICAL TRIAL: NCT04293861
Title: Evaluation of the Evolution of Biological and Imaging Markers of Bone and Cartilage Degradation in Patients With Knee Osteoarthritis Receiving Intra-articular Injections of a Hyaluronan Derivative HYMOVIS®
Acronym: MOKHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EQC5-14-02
Record Dates: First submitted 2020-03-02; First posted 2020-03-03 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Knee Osteoarthritis
Keywords: Hyaluronic acid; MRI; Biomarkers; Cartilage; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HYMOVIS Arm (Experimental): A treatment cycle consists of two injections administered at one week interval. For the purpose of this study, two treatment cycles of two injections of HYMOVIS® at baseline and 6 months will be performed per patient at V1 (Day 0), V2 (Day 7), V5 (Day 180) and V6 (Day 187).
  Interventions: Device: HYMOVIS

INTERVENTIONS:
Device: HYMOVIS — HYMOVIS is a clear hydrogel obtained by hydration of the HA-based derivative named HYADD4p5. The conjugate compound is constituted by a partial hexadecylamide of hyaluronic acid, which is produced by a fermentation process.

SUMMARY:
This pilot study MOKHA is aimed to evaluate the beneficial effect of HYMOVIS® on cartilage of patients suffering of knee osteoarthritis as revealed by using scientifically sound, objective measurements of biological and MRI-based imaging markers.

DETAILED DESCRIPTION:
This study is a post-marketing, open-label, prospective and multicentric pilot study in 50 patients suffering from knee OA. Investigators will be rheumatologists or articular disease specialists from public or academic hospitals located in Belgium and France. In each investigating center, the same injector will perform all the VS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age of 40 and 80 with BMI ≤ 40
* Monolateral (unless contralateral knee is grade I and asymptomatic) femorotibial knee OA associated or not with femoropatellar knee OA

  * Responding to clinical and radiological criteria of the American College of Rheumatology (ACR) (Appendix 1)
  * Symptomatic for more than 6 months in the most painful knee
  * Radiological Kellgren & Lawrence (K&L) II or III in radiographs from less than 12 months (Appendix 2)
* Mean knee pain score at rest over the last 24 hours evaluated on VAS (0-100) ≥ 40 (Appendix 3) with a washout period for Paracetamol and oral NSAIDs depending on the half-life of the drug (Appendix 4). The most painful knee is considered.
* Able to follow the instructions of the study
* Having signed an ICF

Exclusion Criteria:

Related to the OA pathology

* Bilateral (except asymptomatic and grade I) OA of the knee
* Radiological K&L grade I or IV (Appendix 2)
* Chondromatosis or villonodular synovitis of the knee
* Recent trauma (< 1 month) of the knee responsible of the symptomatic knee
* Acute inflammatory OA (KOFUS (Knee Osteoarthritis Flare Up Scale) score ≥ 7, Appendix 5)
* Articular disease resulting from articular dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, hemophilia, hemochromatosis….
* Inflammatory disease i.e. rheumatoid arthritis, gout, infectious arthritis, acute calcium pyrophosphate arthritis
* Pathologies interfering with the evaluation of OA (radiculalgia in the lower limbs, arteritis…..)
* Presence of another joint (other than the target knee) affected by OA (confirmed in radiographs and symptomatic)

Related to treatments

* Corticosteroids injection in the target knee in the last month before first injection
* Hyaluronan injection in the target knee in the last 6 months before first injection
* Arthroscopy and surgery in the target knee in the last 6 months before first injection
* Oral corticotherapy ≥ 5mg/day (in Prednisone equivalent) in the last 3 months before first injection
* OA treatments based on curcuma extract (e.g. FLEXOFYTOL) in the last 3 months before first injection
* Change in the dosage of SYSAD i.e. chondroitin, glucosamine, diacerein or avocado-soy unsaponifiables in the last 3 months before first injection
* Paracetamol and oral NSAIDs before inclusion and follow-up visits (washout period depending on the half-life of the drug, Appendix 4).
* Osteoporosis-related treatments based on strontium ranelate, selective estrogen-receptor modulator (SERM) and parathormone (PTH) in the last 12 months before first injection
* An anticipated need for any forbidden OA treatments during the trial
* Contraindications to HYMOVIS®: hypersensitivity to the product components and infections or skin diseases in the area of the injection site.
* Non-pharmacologic therapy (including physical therapy) for the lower extremities initiated in the month before first injection
* Anticoagulant (coumarinic compound) and heparin

Related to associated diseases

* Severe diseases (liver or renal failure, lung/heart disease, tumor, HIV….)
* Allergy or contra-indication to hyaluronan
* Severe alteration of mobility enabling functional evaluation
* High risk of hemorrhage and risk of infection at the site of injection
* Anticipated need for any surgical or other invasive procedure during the trial including prosthesis in the target knee

Related to patients

* Participation to a therapeutic clinical trial in the last 3 months before first injection
* Under guardianship or judicial protection
* Pregnancy, breastfeeding, planned conception, premenopausal women without contraception, tubal ligation or hysterectomy

Related to MRI counter-indication

* Patient with a pacemaker, an implantable defibrillator, neurosurgical clips, a neurostimulator, cochlear implant, a stent from less than 3 weeks, an insulin pump
* Patient with a ferromagnetic splinter in the body, or having wire sutures
* Serious mobility problem (Parkinson, tremors),
* Claustrophobia

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Assess the variation of type II collagen-specific biomarkers (Coll2-1, Coll2-1NO2 & CTX-II) after HYMOVIS® treatment versus baseline | Variation of levels of biomarkers from baseline (V1) trough 1 year follow up (V8)
  Measure of the level of Coll2-1, Coll2-1NO2 and CTX-II biomarkers in biological fluids.

SECONDARY OUTCOMES:
Variation in biomarkers related to cartilage homeostasis (synthesis/degradation balance) after HYMOVIS® treatment vs. baseline | ariation of levels of biomarkers from baseline (V1) trough 1 year follow up (V8)
  Level of Agrec, COMP, PIIANP, MMP-3 -MPO and IL-6 biomarkers.
Variation in MRI markers after HYMOVIS® treatment vs. baseline | trough 1 year follow up
  Semi-quantitative WORMS - T2 relaxation time (T2 mapping) - Cartilage parameters (volume, thickness, curvature)
Variation in pain and function | trough 1 year follow up
  Pain and function evaluated with KOOS index - VAS for the mean knee pain over the last 24 hours at rest and while walking pain - VAS for global assessment of disease activity (by patient and by investigator)
Responder to treatment | trough 1 year follow up
  Responder rate to treatment (OARSI OMERACT criteria)
Tolerance and satisfaction | trough 1 year follow up
  Adverse events and drop-off - Patient satisfaction scale

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (4):
  - Service de Rhumatologie CHU Dinant-Godinne (Site Godinne), Yvoir, Namur
  - Service de Rhumatologie, CHU Brugmann, Brussels
  - CHR Citadelle de Liège, Liège
  - Service de Rhumatologie CHU Liège, Liège
- France (4):
  - Service de Rhumatologie CHR Metz Thionville Hôpital Bel Air, Thionville, Thionville Cedex
  - Hopital Edouard Herriot (Lyon), Lyon
  - Service de rhumatologie,RDC Hôpital Lariboisière, Paris
  - Centre Hospitalier Nord Franche-Comté, Trévenans